CLINICAL TRIAL: NCT04313959
Title: Comparison of Two Anesthetic Techniques in Blocking the Erector Plane of the Spine Bilateral in Cardiac Surgery: a Prospective Randomized Double-blinded Clinical Trial
Brief Title: Comparison Erect Spine in Cardiac Surgery
Acronym: COESPINE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Coracao (Other Government)
Responsible Party: Principal Investigator, Filomena R B G Galas, Associate Professor of Anesthesiology at University São Paulo Medical School, Instituto do Coracao
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 27166919.3.0000.0068
Record Dates: First submitted 2020-03-17; First posted 2020-03-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Spine Erector; Cardiac Surgery; Acute Pain; Chronic Pain
Keywords: Spine erector; Cardiac surgery; Coronary arterial bypass surgery; Acute Pain; Ropivacaine; Dexamethasone
MeSH Terms: conditions — Acute Pain; Chronic Pain | interventions — Ropivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local anesthetic (Active Comparator): Patients assigned for local anesthetic group will receive a single-shot ultrasound-guided erector spine plane block with 25 mL of 0.2% of ropivacaine
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution
- Local anesthetic + steroid (Active Comparator): Patients assigned for local anesthetic + steroid group will receive a single-shot ultrasound-guided erector spine block plane with 25 mL of 0.2% of ropivacaine with 5 mg dexamethasone
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution; Drug: Ropivacaine 0.2% + Dexamethasone

INTERVENTIONS:
Drug: Ropivacaine 0.2% Injectable Solution — Single-shot ultrasound-guided erector spine plane block of 0.2% ropivacaine
  Other Names: Do not have
Drug: Ropivacaine 0.2% + Dexamethasone — Addiction of 5 mg/ml dexamethasone in 0.2% ropivacaine solution
  Other Names: Do not have
  Arms: Local anesthetic + steroid

SUMMARY:
Open cardiac surgeries are characterized by the increased use of opioids and longer extubation times, being post-sternotomy pain one of the causes of greater patient discomfort, plexus blockages have been used more frequently given the good results of anatomical studies and case series that are just beginning to be published. however, there is not enough data to convince the scientific community of its advantages, continuing to carry out its performance due to lack of evidence. Dexamethasone also shows an excellent result blocking the inflammatory chain and it was evidenced that it prolongs the time of blockages when used perineurally in the plexus blockages. This study wants to show the improvement of pain in patients who undergo this type of surgery and also show the advantages of a longer blockage, which can reduce use of analgesic and opioids, as well as decrease the time of hospitalization This is a double-blinded, randomized, clinical trial designed to determine the efficacy of spine erector whit dexamethasone gives more duration of the blockage and less pain after cardiac surgery.

DETAILED DESCRIPTION:
Evaluation of acute pain pos cardiac surgery in patients that who were subjected at myocardial revascularization. We offer Espine erector block (ESP) with linear array Transducer and needle 100mm bilateral as a technique that offer results more hopeful and less invasive in patients with open cardiac surgery. Favoring the implementation of Fastrack anesthesia techniques in cardiac surgery and minimizing complications in this group of patients

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery bypass graft with cardiopulmonary bypass
* Left ventricular ejection fraction ≥ 45%

Exclusion Criteria:

* Reoperation
* Low cardiac output syndrome
* Preoperative coagulopathy
* Presence of ventricular assist device other than intraaortic ballon pump
* Emergency procedures
* Bacterial or fungal infection in the preceding 30 days
* Active neoplasia
* Allergy or intolerance to steroids
* Allergy to ropivacaine
* Patient refusal
* Participation in other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-02-25 (Estimated); Study Completion 2023-04-17 (Estimated)

PRIMARY OUTCOMES:
Pain intensity score | Within 7 days after cardiac surgery
  Changes in Numeric Rating Scale (NRS) and visual analogue scale (VAS) will be recorded daily at postoperative 1 to 7 day or until the patient's hospital discharge if this occurs before 7 days.
  * Numerical rating scales A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable
  * VAS have also been utilized in EMA research. VAS are measures of subjective or behavioral experience (e.g., pain, physical exercise). They are typically presented as a 10 cm line with descriptive anchors at each end, such as "completed all prescribed activities today" to "completed none of the prescribed activities today." Respondents place a vertical line through the point on the scale that best fits their experience with that construct at that moment.

SECONDARY OUTCOMES:
Total opioids consumption | Up to 2 postoperative day
  The total amount of opioids given by patient
Pain intensity score | Up to 90 days
  Changes inThe Brief Pain Inventory (BPI).will be recorded after discharge at 30 days, 60 days and 90 days after surgery
  *The Brief Pain Inventory (BPI) rapidly assesses the severity of pain and its impact on functioning; BPI Pain Items, Least pain in last 24 hours, Pain on average, Pain right now, Worst pain in last 24 hours; BPI Interference Items, Mood, Walking ability, Normal work (including housework), General activity, Relations with other people, Sleep, Enjoyment of life
Duration of mechanical ventilation | Within 7 days after cardiac surgery
  Duration in hours from the intraoperative intubation up to postoperative extubation

CONTACTS AND LOCATIONS:
Overall Officials: Luis Alberto Rodriguez Linares, MD, Principal Investigator — INCOR FMUSP
Locations (1):
- Incor - Heart Institute - University of Sao Paulo, São Paulo, Brazil